CLINICAL TRIAL: NCT05193526
Title: COronaVirus Induced Acute Respiratory Disease Syndrome During PREGnancy
Acronym: COVADIS-PREG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: COVADIS PREG
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Distress Syndrome Related to SARS-CoV-2
Keywords: COVID-19,; Acute respiratory distress syndrome; Pregnancy; Preterm delivery; SARS-CoV-2; ICU; Critical Care; Mechanical ventilation
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Few data are available on the management of critically ill pregnant women with pneumonia related to SARS-CoV-2. In the absence of clear recommendations for the management of delivery, clinicians are faced with the risk of pregnancy continuation against the risk of premature birth. In these multicenter retrospective study, the investigators want to describe clinicians attitude on delivery management in pregnant women requiring invasive mechanical ventilation for acute respiratory distress syndrome related to SARS-CoV-2.

Two strategies will be compared on maternal, obstetric and neonatal outcomes:

* Wait strategy defined by no extraction within 24 hours of invasive venting
* Early strategy defined by extraction within 24 hours of invasive ventin

ELIGIBILITY:
1. patient > 18 years
2. Patient with SARS-CoV-2 pneumonia proven by RT-PCR
3. Hospitalization in an intensive care unit during pregnancy after 14 weeks' gestation
4. Need for ventilatory support including: oxygen therapy > 6L/min and/or NIV and/or High Flow Oxygen and/or invasive mechanical ventilation +/- ECMO.

Exclusion Criteria:

* Patient's refusal to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women after 14 week of amenorrhoea with SARS-CoV-2 pneumonia requiring ICU admission for acute respiratory distress syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Compare two fetal extraction strategies: - Wait strategy defined by no extraction within 24 hours of invasive venting - Early strategy defined by extraction within 24 hours of invasive venting | 'Day 1.
  Assessment Criterion 1: Maternal prognosis assessed by:
  * Mortality
  * Duration of invasive mechanical ventilation
  * Need for ECMO
  * Use of prone position and/or nitric oxide and/or almitrine
  * Adverse events: cardiac arrest, organ failure, thromboembolic episodes, nosocomial infections, barotrauma
  * Length of stay in the ICU and in the hospital
  Assessment Criterion 2: Obstetric prognosis assessed by:
  * Fetal extraction in the ICU room due to a contraindication to transport (maternal and/or fetal risk)
  * Delivery route
  * Peri partum hemorrhage
  * Complications of obstetric anesthesias
  Assessment Criterion #3: Fetal Prognosis Assessed by:
  * Term birth,
  * Weight,
  * Apgar,
  * pH cord blood,
  * Need for ICU admission,
  * Death

SECONDARY OUTCOMES:
Number of patient requiring invasive mechanical ventilation with or without ECMO | 'Day 1.
  Number of patient requiring invasive mechanical ventilation with or without ECMO
Number of patients receiving pharmacological treatments for the management of COVID: corticosteroids, antivirals, anti-IL6, anticoagulants, antibiotics | Day 1.
  Number of patients receiving pharmacological treatments for the management of COVID: corticosteroids, antivirals, anti-IL6, anticoagulants, antibiotics
Evolution over time of the number of patients admitted to the ICU in the participating | Day 1.
  Evolution over time of the number of patients admitted to the ICU in the participating centers (1st, 2nd, 3rd epidemic wave)
Evolution over time of the number of patients admitted to the ICU in the participating | Day 1.
  Evolution over time of the number of patients admitted to the ICU in the participating

CONTACTS AND LOCATIONS:
Overall Officials: Frederique SCHORTGEN, PhD, Principal Investigator — Centre Hospitalier Intercommunal Créteil
Locations (1):
- 40 Avenue de Verdun, Créteil, France

REFERENCES:
- [Derived] Schortgen F, Tabra Osorio C, Demiri S, Dzogang C, Jung C, Lavenu A, Lecarpentier E; COVADIS-PREG study group. Management of pregnant women in tertiary maternity hospitals in the Paris area referred to the intensive care unit for acute hypoxaemic respiratory failure related to SARS-CoV-2: which practices for which outcomes? Ann Intensive Care. 2024 Jun 18;14(1):94. doi: 10.1186/s13613-024-01313-2. PMID 38890164